CLINICAL TRIAL: NCT00001003
Title: Aerosols in the Treatment of Pneumocystis Carinii Pneumonia: A Nested Study Quantitating the Delivery of Aerosolized Pentamidine for Prophylaxis of PCP in Protocols ACTG 021 and ACTG 081
Brief Title: A Study of Pentamidine in the Prevention of Pneumocystis Carinii Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 079; 11054 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Nebulizers and Vaporizers; Lung; Administration, Inhalation; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Respiratory Aspiration; Acquired Immunodeficiency Syndrome | interventions — Pentamidine; Zidovudine

INTERVENTIONS:
Drug: Pentamidine isethionate
Drug: Zidovudine

SUMMARY:
To evaluate and compare 3 anti-pneumocystis regimens plus zidovudine (AZT) in persons with advanced HIV disease and T4 cell count < 200 cells/mm3. To establish the range of pentamidine (PEN) deposition in AIDS patients participating in ACTG 021 and ACTG 081. To identify factors (breathing pattern, pulmonary function) that may be important in affecting the actual dose delivered to a given patient.

The specific system that is used to deliver PEN to the lungs may determine whether a therapeutically effective dose is attained in the lungs. Therefore, this study will establish the amount of PEN that is deposited in the lungs of patients enrolled in protocols ACTG 021 and ACTG 081, who are being treated with PEN administered from the Marquest Respirgard II nebulizer.

DETAILED DESCRIPTION:
The specific system that is used to deliver PEN to the lungs may determine whether a therapeutically effective dose is attained in the lungs. Therefore, this study will establish the amount of PEN that is deposited in the lungs of patients enrolled in protocols ACTG 021 and ACTG 081, who are being treated with PEN administered from the Marquest Respirgard II nebulizer.

Approximately 4 weeks after patients in ACTG 021 and ACTG 081 have begun PEN aerosol therapy for the prevention of PCP, patients undergo the first radioactive aerosol study. The patient inhales a mist while sitting with his/her back against a gamma camera. The resulting picture outlines the lungs. This mist contains a single dose of PEN mixed with a small amount of radioactivity (99m-technetium ertechnetate). The gamma camera determines where the particles deposit in the lungs. The radioactivity exposure is equivalent to a typical xray of the ribs. This procedure takes about 45 minutes; 6 hours later another 30-minute gamma camera image is obtained. Blood is withdrawn to measure the blood level of PEN as done in ACTG 021 and ACTG 081. The entire procedure is repeated near the end of the prophylactic schedule (about 10-12 months after the start of aerosol PEN treatments).

ELIGIBILITY:
Inclusion Criteria

Concurrent Treatment:

Allowed:

* Local radiation for Kaposi's sarcoma.

Patients who successfully completed a course of study therapy for acute Pneumocystis carinii pneumonia (PCP) and who met the inclusion criteria for Protocol ACTG 021 or ACTG 081 and were randomized to the aerosolized pentamidine arm.

* Patients who are currently receiving aerosolized pentamidine as prophylactic therapy for PCP.

Exclusion Criteria

The following patients are excluded:

* Those enrolled in ACTG 021 and randomized to the oral prophylaxis arm.
* Those enrolled in ACTG 081 and randomized to the trimethoprim / sulfamethoxazole and dapsone arms.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Transfusions of blood or red blood cells.

Co-Existing Condition:

* Significant adverse effects.

Active substance abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Study Completion 1992-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GC Smaldone, Study Chair
Locations (1):
- SUNY - Stony Brook, Stony Brook, New York, United States

REFERENCES:
- [Background] Smaldone GC, Fuhrer J, Steigbigel RT, McPeck M. Factors determining pulmonary deposition of aerosolized pentamidine in patients with human immunodeficiency virus infection. Am Rev Respir Dis. 1991 Apr;143(4 Pt 1):727-37. doi: 10.1164/ajrccm/143.4_Pt_1.727. PMID 2008984